CLINICAL TRIAL: NCT00187291
Title: Alternans Before Cardioverter Defibrillator (ABCD) Trial
Brief Title: Study to Compare TWA Test and EPS Test for Predicting Patients at Risk for Life-threatening Heart Rhythms (ABCD Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Cambridge Heart Inc. (Industry); MetroHealth Medical Center (Other)
Responsible Party: David Rosenbaum, MD, MetroHealth Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: G010050
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Cardiomyopathy; LV Dysfunction
Keywords: T-Wave Alternans; ICD; Primary Prevention
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: T-Wave Alternans test

SUMMARY:
The ABCD clinical study is designed to determine if a T-Wave Alternans (TWA) test is equivalent to an Electrophysiology Study (EPS) in predicting life-threatening heart rhythms in patients with ischemic heart disease, left ventricular dysfunction, and non-sustained tachycardia. Patients undergo both the TWA test and EP study and receive an Implantable Cardioverter Defibrillator (ICD)if either of the tests show the patient is at risk. The patient is then followed for 2 years. The incidence of a ventricular tachyarrhythmia events and total mortality are to be evaluated over the duration of the study.

DETAILED DESCRIPTION:
The primary objective of this study is to test the hypothesis that therapy directed primarily by a T wave alternans (TWA) test, measured non-invasively during exercise, is equivalent to therapy directed by an electrophysiological study (EPS) in predicting spontaneous ventricular tachyarrhythmic events (VTEs) in patients with ischemic heart disease, left ventricular dysfunction, and asymptomatic non-sustained ventricular tachycardia (NSVT).

In the absence of any previous life-threatening ventricular arrhythmia (i.e., for primary prevention), ICD implantation is currently indicated in patients with ischemic heart disease, left ventricular dysfunction, asymptomatic non-sustained ventricular tachycardia, and a positive EPS. The objective of this study is to demonstrate that a TWA test directed therapy is equivalent to EPS directed therapy in guiding ICD implantation for the purpose of primary prevention of sudden cardiac death (SCD) in patients with ischemic heart disease, left ventricular dysfunction, and asymptomatic non-sustained ventricular tachycardia.

This is a prospective, multi-center study to demonstrate the following:

PRIMARY HYPOTHESIS: a TWA test directed therapy is equivalent to EPS directed therapy in predicting VTEs in patients with ischemic heart disease, LVEF less than 0.40, and asymptomatic non-sustained ventricular tachycardia. The study will determine whether the positive predictive value of TWA test directed therapy is equivalent to the positive predictive value of EPS directed therapy. The study will also determine whether the negative predictive value of TWA test directed therapy is equivalent to the negative predictive value of EPS directed therapy. The positive groups under TWA test directed therapy will be compared with the positive groups under EPS directed therapy, and the negative groups under TWA directed therapy will be compared with the negative groups under EPS directed therapy. SECONDARY HYPOTHESIS: The study will determine whether the positive predictive value of a TWA test (not including indeterminates) is equivalent to the positive predictive value of an EPS in predicting future VTEs. The study will also determine whether the negative predictive value of a TWA test (not including indeterminates) is equivalent to the negative predictive value of an EPS in predicting future VTEs. The TWA test positive groups will be compared with the EPS positive groups, and the TWA test negative groups will be compared with the EPS negative groups. The secondary hypothesis will also be tested against the primary endpoint defined above.

ELIGIBILITY:
Inclusion Criteria:

Patients with no previous history of life threatening ventricular arrhythmias or symptomatic non-sustained VT, and who meet the following inclusion criteria may be enrolled in the study:

1. Ischemic heart disease as documented by any of the following: previous myocardial infarction (documented by 2 out of 3 of the following: history, ECG, and/or cardiac enzymes), prior PTCA or CABG; angina with a positive exercise or pharmacological stress test; angina with a greater than 50% occlusion of any coronary artery, left ventricular dysfunction that can be attributed to angiographically documented coronary artery disease
2. LVEF less than 0.40 as determined by echocardiography, radionuclide or contrast ventriculography within six months of enrollment.
3. Non-sustained ventricular tachycardia within 6 months of enrollment, defined as greater than 3 consecutive premature ventricular contractions having at least three consecutive intervals with a cycle length at or below 550 ms, and with the entire episode lasting less than 30 seconds. This episode should be associated with either no symptoms, or palpitations alone. An episode of NSVT associated with any symptoms (other than palpitations) does not satisfy inclusion criteria for the trial.
4. The patient is 18 years of age or older.
5. In the judgement of the principal investigator, the patient is capable of undergoing a sub-maximal treadmill exercise test to a heart rate of 120 bpm.
6. The patient has signed the latest IRB approved informed consent form.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria will not be eligible for enrollment:

1. The patient is unable to give informed consent.
2. The patient is known to have had a cardiac arrest or sustained life threatening ventricular arrhythmias, other than in the setting of an acutely reversible cause (e.g., acute phase MI, drug intoxication).
3. The patient has had an EPS or TWA test at any time and for any reason prior to being screened and consented for this trial.
4. The patient has unstable coronary artery disease.
5. The patient has contraindications to ICD implantation.
6. A submaximal exercise test is contraindicated.
7. The patient has persistent atrial fibrillation or flutter.
8. The patient is less than 28 days post MI, post CABG, or post coronary angioplasty.
9. The patient has an LVEF 0.40, but no evidence of ischemic heart disease as defined by section 4.1.
10. The patient has NYHA functional Class IV congestive heart failure symptoms at the time of enrollment.
11. The patient is on any class 1 or 3 antiarrhythmic drug.
12. The patient is participating in a study of another investigational device or drug. If, in the opinion of the investigator, this would not interfere with this study, the eligibility of such a patient should be discussed with the primary investigators of the ABCD trial, Drs. Rosenbaum or Costantini.
13. The patient has any other significant medical condition or acute illness that in the opinion of the investigator precludes participation.
14. The patient has a previous history of syncope, unless the episode was clearly not caused by a ventricular tachyarrhythmia.
15. The patient has a life expectancy of less than one year from any cause.
16. The patient has a positive pregnancy test.
17. The patient is not geographically stable or is unable to comply with the follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618
Dates: Start 2001-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Ventricular tachyarrhythmic events | 12 months

SECONDARY OUTCOMES:
Total Mortality | 12 months
Ventricular tachyarrhythmic events below rate detection of the ICD | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenbaum, MD, Study Chair — MetroHealth Medical Center; Otto Costantini, MD, Study Chair — MetroHealth Medical Center

REFERENCES:
- [Derived] Costantini O, Hohnloser SH, Kirk MM, Lerman BB, Baker JH 2nd, Sethuraman B, Dettmer MM, Rosenbaum DS; ABCD Trial Investigators. The ABCD (Alternans Before Cardioverter Defibrillator) Trial: strategies using T-wave alternans to improve efficiency of sudden cardiac death prevention. J Am Coll Cardiol. 2009 Feb 10;53(6):471-9. doi: 10.1016/j.jacc.2008.08.077. PMID 19195603